CLINICAL TRIAL: NCT03611322
Title: A Trial to Compare Pharmacokinetic Properties of Semaglutide Following Subcutaneous Administration of Semaglutide 1 mg by the DV3372 Device and by the PDS290 Semaglutide Pen-injector
Brief Title: A Trial to Compare Blood Concentration Levels of Semaglutide Following Subcutaneous Injections of Semaglutide 1 mg by 2 Different Devices (the DV3372 Device and by the PDS290 Semaglutide Pen-injector)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4429; U1111-1206-9372 (Other: World Health Organization (WHO)); 2017-005127-25 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DV3372 device (Experimental): Participants will receive semaglutide on day 1, 8, 15, 22 and 29. The treatment period from first treatment (Day 1) to end of the treatment (Day 29) will be 4 weeks.
  Interventions: Drug: Semaglutide, 0.25 mg; Drug: Semaglutide, 0.5 mg; Drug: Semaglutide, 1.0 mg; Device: DV3372
- PDS290 semaglutide pen-injector (Active Comparator): Participants will receive semaglutide on day 1, 8, 15, 22 and 29. The treatment period from first treatment (Day 1) to end of the treatment (Day 29) will be 4 weeks.
  Interventions: Drug: Semaglutide, 0.25 mg; Drug: Semaglutide, 0.5 mg; Drug: Semaglutide, 1.0 mg; Device: PDS290 pen-injector

INTERVENTIONS:
Drug: Semaglutide, 0.25 mg — Semaglutide will be administered subcutaneously (s.c., under the skin) on day 1 and 8 in the morning after an overnight fast of at least 8 hours
Drug: Semaglutide, 0.5 mg — Semaglutide will be administered s.c. (under the skin) on day 15 and 22 in the morning after an overnight fast of at least 8 hours
Drug: Semaglutide, 1.0 mg — Semaglutide will be administered s.c. (under the skin) on day 29 in the morning after an overnight fast of at least 8 hours
Device: DV3372 — DV3372 device will be used for administration of semaglutide
  Arms: DV3372 device
Device: PDS290 pen-injector — PDS290 pen-injector will be used for administration of semaglutide
  Arms: PDS290 semaglutide pen-injector

SUMMARY:
This study compares semaglutide in two different injection tools called "PDS290" and "DV3372". The study aims to show similar levels of semaglutide in the blood when using either of the two injection tools. The researchers also want to look at how well the injection tools work. Participants will either receive semaglutide using the PDS290 or the DV3372 injection tool. This is decided by chance, like flipping a coin. This is called randomisation. Semaglutide is an approved medicine (thus available on the market) for people with type 2 diabetes. Semaglutide will be injected subcutaneously (injection under the skin). Participants will get a total of 5 injections with semaglutide. The study will last for a maximum of 86 days. Participants will have 17 scheduled site visits with the study physician or study staff at the study centre. For one of the visits participants will stay at the research unit for 4 days and 3 nights. Participants cannot take part in this study if participants have any disorder that the doctor thinks is a health problem. Only healthy men and women are allowed to take part. Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria: - Male or female, aged 18 to 55 years (both inclusive) at the time of signing informed consent. - Body mass index between 20.0 and 29.9 kg/m^2 (both inclusive) and weight between 55.0 and 90.0 kg (both inclusive). - Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator. Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive methods. - Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol. - Use of prescription medicinal products or non-prescription drugs or herbal products, except routine vitamins, topical medication, highly effective contraceptives and occasional use of paracetamol (not allowed within 24 hours before screening), within 14 days prior to the day of screening. - Abuse or intake of alcohol, defined as any of the below: 1) Known or suspected alcohol abuse within 1 year prior to the day of screening (defined as regular intake of more than an average intake of 24 g alcohol daily for men and 12 g alcohol daily for women -12 g of alcohol equals about 300 mL of beer or lager, 100 mL of wine, or 25 mL spirits) or 2) Positive alcohol test at screening. - Abuse or intake of drugs, defined as any of the below: 1) Known or suspected drug/chemical substance abuse within 1 year prior to the day of screening or 2) Positive drug of abuse test at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
AUC0-last,sema,Week5: the area under the plasma semaglutide concentration-time curve from 0 until last quantifiable measurement after first maintenance dose of subcutaneous semaglutide 1 mg administration following a four week escalation period | 0-840 hours (5 weeks)
  Measured in nmol*h/L
Cmax,sema,Week5: the maximum plasma semaglutide concentration after first maintenance dose of subcutaneous semaglutide 1 mg administration following a four week escalation period | 0-840 hours (5 weeks)
  Measured in nmol/L

SECONDARY OUTCOMES:
tmax,sema,Week5: time to Cmax of semaglutide after first maintenance dose of subcutaneous semaglutide 1 mg administration following a four week escalation period | 0-840 hours (5 weeks)
  Measured in hours
t½,sema,Week5: terminal elimination half-life of semaglutide after first maintenance dose of subcutaneous semaglutide 1 mg administration following a four week escalation period | 0-840 hours (5 weeks)
  Measured in hours
Number of site-initiated technical complaints with or without co-reported adverse events | from first semaglutide dose (day 1) and until the follow-up visit (5 weeks after the last dose of semaglutide)
  Number of technical complaints

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com